CLINICAL TRIAL: NCT04029519
Title: A Multicenter, Open-Label Retreatment Study of the Safety and Effectiveness of PN40082 for Lip Augmentation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Prollenium Medical Technologies Inc. (Industry)
Collaborators: Symbio, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO 2018-03
Record Dates: First submitted 2019-07-18; First posted 2019-07-23 (Actual); Results first posted 2021-07-14 (Actual); Last update posted 2021-07-14 (Actual); Status verified 2021-06

CONDITIONS: Lip Augmentation

STUDY DESIGN:
Intervention Model Description: multicenter, open-label clinical study of retreatment of subjects seeking lip augmentation
Masking Description: Open Label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- PN40082 (Experimental): All subjects in this study will receive one open-label treatment with PN40082.
  Interventions: Device: PN40082

INTERVENTIONS:
Device: PN40082 — PN40082 (manufactured by Prollenium Medical Technologies) is a clear, colorless gel in 1.0 mL pre-filled syringes with 25 mg/mL of stabilized hyaluronic acid and lidocaine 0.3% w/w.

SUMMARY:
To evaluate the safety and efficacy of retreatment with PN40082 for lip augmentation.

DETAILED DESCRIPTION:
This is a multicenter, open-label clinical study of retreatment of subjects seeking lip augmentation who received treatment with either PN40082 or Restylane Silk in prior Protocol PRO 2018-02 (NCT04032977). Subjects meeting the inclusion/exclusion criteria will receive a single additional treatment with PN40082

ELIGIBILITY:
Inclusion Criteria:

1. In Protocol PRO 2018-02, the subject was in the per-protocol population, i.e., met all inclusion/exclusion criteria; received study device, completed Visit 5 within the specified window; had LFGS score by the Blinded Evaluating Investigator at Visit 3/Month 2, and had no significant protocol violations that would affect the treatment evaluation.
2. If female and of childbearing potential, a negative urine pregnancy test at Visit 1/Day 1 and the subject agrees to use adequate contraception during the study period
3. Willing to give written informed consent

Exclusion Criteria:

1. Women who are pregnant, lactating, or planning a pregnancy

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2018-12-21 (Actual); Primary Completion 2019-08-27 (Actual); Study Completion 2019-08-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stacy R. Smith, MD, Principal Investigator — California Dermatology & Clinical Research Institute
Locations (6):
- United States (6):
  - California Dermatology & Clinical Research Institute, Encinitas, California
  - International Dermatology Research, Inc, Miami, Florida
  - Skin Specialists, PC, Omaha, Nebraska
  - Schweiger Dermatology, PLLC, New York, New York
  - Tennessee Clinical Research Center, Nashville, Tennessee
  - Skintastic, Plano, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | PN40082
Started | 84
Completed | 79
Not Completed | 5
Not completed — Protocol Violation | 1
Not completed — Withdrawal by Subject | 3
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | PN40082
Number analyzed (Participants) | 84
Age, Continuous [Mean (Full Range); unit: years] | 50 [24 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 82
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17
  Not Hispanic or Latino | 67
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 12
  White | 70
  More than one race | 1
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Lip Fullness Grading Scale
Description: Lip Fullness Grading Scale is a validated 5-point photonumeric rating scale with 0 being very thin lips (worse outcome) up to 4 full lips (best outcome)
Time Frame: Visit 1/Day 1 to Visit 3/Month 2, 56 Days
Population: Change from Baseline in Overall Lips Fullness Grading Scale at Visit3/Month 2.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PN40082
Number analyzed (Participants) | 79
score on a scale | .82 (0.747)

2. Primary Outcome: Change From Baseline in Perioral Lines Severity Scale
Description: Change from baseline in the perioral lines rating scale (POL), a 4 point rating scale with 0 as a mouth with no perioral lines (better outcome) to 3 a mouth with many deep lines or crevices (worse outcome).
Time Frame: Visit 1/Day 1 to Visit 3/Month 2, 56 Days
Population: Change from baseline to Visit 3/Month 2 in the perioral lines rating scale for the 17 subjects who had perioral lines treated.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PN40082
Number analyzed (Participants) | 17
score on a scale | -0.75 (0.577)

3. Secondary Outcome: Number of Participants With Patient Global Aesthetic Improvement
Description: Change from baseline for the patient Global Aesthetic Improvement scale, a 5 point scale with 1= the appearance is worse than the original condition (worse outcome) up to 5 very much improved optimal cosmetic result (better outcome)
Time Frame: Visit 1/Day 1 to Visit 3/Month 2, 56 days
Population: Change from baseline in the Patient Global Aesthetic Improvement scale with 5 being much improved optimal cosmetic results (better outcome) and 1 being the appearance is worse than the original condition (worse outcome)
Measure: Count of Participants; unit: Participants
Arm/Group | PN40082
Number analyzed (Participants) | 79
Participants
  Very much Improved (5) | 41
  Much Improved (4) | 19
  Improved (3) | 17
  No change (2) | 2
  Worse (1) | 0

4. Secondary Outcome: Number of Participants With Investigator Global Aesthetic Improvement
Description: Change from baseline in the Investigator Global Aesthetic Improvement score, a 5 point scale with 1= the appearance is worse than the original condition (worse outcome) up to 5 = very much improved optimal cosmetic result (better outcome)
Time Frame: Visit 1/Day 1 to Visit 3/Month 2, 56 days
Population: Change from baseline in the Investigator Global Aesthetic Improvement score with 1 being appearance is worse than the original condition (worse outcome) up to 5 being very much improved optimal cosmetic result (better outcome)
Measure: Count of Participants; unit: Participants
Arm/Group | PN40082
Number analyzed (Participants) | 79
Participants
  Very Much Improved (5) | 28
  Much Improved (4) | 30
  Improved (3) | 20
  No Change (2) | 1
  Worse (1) | 0

5. Secondary Outcome: Number of Subjects With Decreased Swelling
Description: Swelling Assessment at Visit 3/Month 2, a 4 point scale with 0 = no swelling (better outcome) up to 4= Severe Swelling (worse outcome)
Time Frame: Visit 1/Day 1 to Visit 3/Month 2, 56 days
Population: Swelling assessment at Visit 3/Month 2 with 0 = no swelling (better outcome) up to 4 = severe swelling (worse outcome)
Measure: Count of Participants; unit: Participants
Arm/Group | PN40082
Number analyzed (Participants) | 79
Participants | 79

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time the subject signed informed consent until discharged from the study, approximately 3 months. Follow-up procedures related to pregnancy, AEs, SAEs or AESIs could continue beyond the end of the study, an average of 6 months.
Arm/Group | PN40082
All-Cause Mortality (participants affected / at risk) | 0/84
Serious Adverse Events (participants affected / at risk) | 1/84
Other Adverse Events (participants affected / at risk) | 61/84
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PN40082 (N=84)
Beta Hemolytic Streptococcal Infection (Infections and infestations) | 1 (2)
Stenosis in Sigmoid Colon (Gastrointestinal disorders) | 1 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PN40082 (N=84)
Injection Site Bruising (General disorders) | 40 (40)
Injection Site Erythema (General disorders) | 6 (6)
Injection site mass (General disorders) | 6 (6)
Injection site pain (General disorders) | 10 (10)
Injection Site Swelling (General disorders) | 48 (48)
Facial Asymmetry (Musculoskeletal and connective tissue disorders) | 5 (5)

LIMITATIONS AND CAVEATS:
There were no limitations of the trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-11-13): https://cdn.clinicaltrials.gov/large-docs/19/NCT04029519/Prot_002.pdf
  • Statistical Analysis Plan (2019-03-06): https://cdn.clinicaltrials.gov/large-docs/19/NCT04029519/SAP_003.pdf